CLINICAL TRIAL: NCT00453089
Title: A Phase I/II Dose Escalation Clinical Trial to Assess Safety and Efficacy of VG101 to Treat the Symptoms of Vulvar and Vaginal Atrophy in Post-Menopausal Women
Brief Title: VG101 Phase I/II to Treat Vulvar and Vaginal Atrophy in Post-Menopausal Women
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bionovo (Industry)
Responsible Party: Mary Tagliaferri, MD, Bionovo, Inc
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VG-101-001
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Vaginal Atrophy; Vulvar Atrophy
Keywords: Chinese Herbs; Postmenopausal; Vaginal Atrophy; Vulvar Atrophy; Symptoms; Bionovo; VG101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: VG101

SUMMARY:
To conduct a prospective, randomized, blinded, placebo controlled, dose escalation clinical trial in 4 cohorts of 10 postmenopausal women (total N=40) aged 45 to 65 years with at least one menopausal vaginal symptom, vaginal pH > 5.0 and > 20% parabasal vaginal epithelial cells.

DETAILED DESCRIPTION:
Primary Aims:

1. the optimal dose of VG101 based on the highest of 4 proposed dose levels that is not associated with unacceptable toxicity during 12 weeks of treatment. Toxicity will be based on National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 3. Unacceptable toxicity will be defined as the occurrence of any Grade 3, 4, of 5 toxicity that is possibly or probably associated with study drug or any other unacceptable toxicity as determined by the Data and Safety Monitoring Board.
2. Specific potential adverse effects of VG101

Secondary Aims:

1. the preliminary efficacy of VG101 to:

   * relieve vulvar and/or vaginal dryness,
   * relieve vulvar and/or vaginal irritation
   * relieve vulvar and/or vaginal itching
   * relieve vulvar and/or vaginal discharge
   * relieve dyspareunia
   * improve sexual function
   * relieve dysuria
   * reduce frequency of urinary incontinence
   * improve quality of life
   * improve the physical examination assessment of vaginal atrophy
   * reduce vaginal fluid pH
   * improve the proportion of superficial vaginal epithelial cells
2. participant adherence to VG101 administration

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 45 and 65
2. Postmenopausal documented by: (a) at least one year of amenorrhea; (b) 6- 12 months of amenorrhea with serum FSH > 40 IU/ml; (c) 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy, or (d) hysterectomy with serum FSH levels > 40 IU/ml.
3. Self-report at least one moderate to severe symptom of vulvar or vaginal atrophy from the following list:

   * Vaginal dryness (none, mild, moderate or severe)
   * Vaginal and/or vulvar discomfort (none, mild, moderate, severe)
   * Vaginal and/or vulvar irritation (none, mild, moderate, severe)
   * Vaginal itching (none, mild, moderate, severe)
   * Vaginal pain associated with sexual activity (none, mild, moderate or severe)
4. < 5% superficial cells on vaginal cytologic smear.
5. Vaginal pH >5.0
6. Willing to use an intravaginal cream containing Chinese herbs for the treatment of vaginal symptoms.
7. Provide informed consent.

Exclusion Criteria:

1. History of breast, uterine or ovarian cancer or melanoma.
2. Abnormal mammogram or breast examination within the last 9 months suggestive of cancer.
3. Abnormal Pap smear or pelvic examination within the last 9 months suggestive of cancer.
4. Any uterine or vaginal bleeding within the six months prior to enrollment (except following the screening Pap smear).
5. Double-wall endometrial thickness that exceeds 5 mm measured on transvaginal ultrasound.
6. Pregnant or lactating.
7. Use of any vaginal moisturizer (Replens, KY Silk-E, Astroglide Silken Secret, Senselle) within 30 days of screening.
8. Use of any oral, transdermal, vaginal, or systemic estrogen or estrogen/progestin product within 30 days of screening.
9. Use of raloxifene, tamoxifen or aromatase inhibitors within 12 weeks of screening.
10. Current urinary tract infection (dipstick urinalysis positive for leukocyte estrace, nitrates or blood)
11. History of cardiovascular disease.
12. History of venous thromboembolic disease.
13. Use of another investigational agent within 12 weeks of screening.
14. Any medical or psychiatric condition that, in the investigator's opinion, would preclude the participant from completing questionnaires or measures, adhering to the protocol or completing the trial, including limited English literacy, severe illness, plans to move, substance abuse, significant psychiatric problems, or dementia.
15. No access to a telephone

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported symptoms of vaginal atrophy from baseline to 12 weeks | 4 and 12 weeks
Change in percent superficial vaginal epithelial cells from baseline 12 weeks | 4 and 12 weeks
Change in the pH of vaginal secretions from baseline to 12 weeks | 4 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary Tagliaferri, MD, Principal Investigator — Bionovo, Inc
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California